CLINICAL TRIAL: NCT04171518
Title: A Real-World Evidence Study in China Boao Lecheng International Medical Tourism Pilot Zone of the Catalys Precision Laser System (Model: Catalys Precision Laser System)
Brief Title: A Real-World Evidence Study in China of the Catalys Precision Laser System
Status: Completed | Type: Observational
Sponsor: Johnson & Johnson Surgical Vision, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CAST-102-SYST
Record Dates: First submitted 2019-11-19; First posted 2019-11-21 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Catalys Precision Laser System: Cataract Surgery with use of Catalys Precision Laser System
  Interventions: Device: Catalys Precision Laser System

INTERVENTIONS:
Device: Catalys Precision Laser System — Cataract surgeons to create a precise anterior capsulotomy and/or subsequent fragmentation (phacofragmentation) of the crystalline lens using the Catalys Precision Laser System

SUMMARY:
This study is a prospective, single-arm, observational study of the Catalys Precision Laser System in real-world clinical practice. The study will be conducted at one site at the Boao Super Hospital in Lecheng International Medical Tourism Pilot Zone of Hainan province in China. The study is being conducted to evaluate the overall performance of the Catalys Precision Laser System. One or both eyes of each subject will be included in study.

The Catalys system is used as part of cataract surgery to create LASER cuts as intended by the surgeon to aid in cataract surgery, without adversely impacting the risk to the patient.As such, the endpoints of surgeon rating of completeness of corneal incisions, anterior capsulotomy and phacofragmentation and any device related adverse events from the time of Catalys System use to 1-month postoperative follow-up should adequately cover the evaluation of the intended use of the Catalys System.

ELIGIBILITY:
Inclusion Criteria

All criteria apply to each study eye:

Note: Study inclusion and exclusion criteria will be per the Catalys system instructions for use. A few key criteria are listed below:

* Patients scheduled for cataract surgery, including treatment with the Catalys Precision Laser System for anterior capsulotomy, phacofragmentation and the creation of single plane and multi-plane arc cuts/incisions in the cornea.
* Signed informed consent and privacy protection authorization or equivalent documentation necessary to comply with applicable privacy laws pertaining to medical treatment and/or medical record in the governing countries
* At least 22 years of age at the time of consent.ion Criteria

Exclusion Criteria:

All criteria apply to each study eye:

* Presence of corneal ring and/or inlay implant(s), Descemetocele with impending corneal rupture)
* Severe corneal opacities, corneal abnormalities, significant corneal edema, or diminished aqueous clarity that obscures OCT imaging of the anterior lens capsule.
* Any contraindications to cataract surgery

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will include subjects undergoing primary cataract extraction and IOL implantation and who meet all the study inclusion and exclusion criteria. Subjects treated during the period of November 2019 to March 2020 (that satisfy the protocol inclusion and exclusion criteria) may be included in the study, or a maximum of 163 subjects (not including the subjects for surgeon certification), whichever comes first. One or both eyes of each subject will be included in study.
Sampling Method: Non-Probability Sample
Enrollment: 139 (Actual)
Dates: Start 2019-11-22 (Actual); Primary Completion 2020-10-12 (Actual); Study Completion 2020-10-12 (Actual)

PRIMARY OUTCOMES:
Rate of successful anterior capsulotomy | Intraoperatively
  If the investigator is able to remove the capsular disc from the peripheral capsule without the need of manual separation of residual tags, then it will be considered a complete capsulotomy.
Rate of successful corneal Incisions | Intraoperatively
  If the investigator is able to blunt dissect the primary incision (without the need for a secondary cutting instrument), then it will be considered a complete cut.
Rate of successful phacofragmentation as intended | Intraoperatively
  If there are no error messages or treatment interruptions occur, then phacofragmentation will be considered complete.

CONTACTS AND LOCATIONS:
Overall Officials: Sanjeev Kasthurirangan, Ph.D., Study Director — Johnson & Johnson Surgical Vision
Locations (1):
- Hainan BoAo Super Hospital, BoAo, Hainan, China

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Devices Companies have an agreement with the Yale Open Data Access (YODA) Project to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA project site at http://yoda.yale.edu
URL: http://yoda.yale.edu